CLINICAL TRIAL: NCT04743856
Title: Advancement of Clinical Referral to Physical Activity for Cardiometabolic Disease Prevention
Brief Title: The Clinical Referral to Activity Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Bonny Rockette-Wagner, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY20030079; 1K01HL151668-01 (NIH)
Record Dates: First submitted 2021-01-10; First posted 2021-02-08 (Actual); Results first posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Physical Inactivity; Cardiovascular Risk Factor; Obesity; Blood Pressure; PreDiabetes
Keywords: Physical activity; Online lifestyle Intervention; Cardiovascular disease; Disease prevention
MeSH Terms: conditions — Sedentary Behavior; Obesity; Prediabetic State; Motor Activity; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 to one of two intervention conditions.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Referring doctors and outcome assessors will be blinded to participant assignment while the study is active. After data collection ends, referring physicians will be informed as to each of their patients assignment. Outcome assessors will remain blinded to participant assignment. Investigators will be blinded to assignment as much as possible. However, certain events ( such as an adverse event report) may cause the study PI to become unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PAT (Physical activity monitor) (Active Comparator): Participants will receive a physical activity tracker and encouragement to increase physical activity.
  Interventions: Behavioral: PAT
- ActiveGOALSv2 (Experimental): Participants will receive the ActiveGOALS online program with an integrated activity tracker.
  Interventions: Behavioral: ActiveGOALSv2

INTERVENTIONS:
Behavioral: ActiveGOALSv2 — 13 weekly self-guided sessions on problem solving and goal setting related to increasing physical activity, and weekly remote coaching support. Once a month support materials sent monthly from months 4-12 of intervention.
  Arms: ActiveGOALSv2
Behavioral: PAT — Participants will receive a physical activity tracker and encouragement to increase activity.
  Arms: PAT (Physical activity monitor)

SUMMARY:
The main aim of this effort is to test a physical activity intervention, for adult clinical care patients at risk of developing cardiovascular disease. The intervention includes social-cognitive theory-based sessions, remote coaching, a body worn physical activity tracker (PAT), and is delivered online over one year. The investigators hypothesis that this intervention will be more successful at increasing physical activity (defined as objectively measured step counts and % of individuals meeting the moderate-vigorous physical activity goal) as an active control group who receives a body worn PAT and information on the CDC activity recommendations. The proposed intervention will be aligned with efforts by the US Centers for Disease Control to increase population physical activity levels and the American College of Sports Medicine (ACSM) to increase physical activity prescription in primary care.

DETAILED DESCRIPTION:
The main aim of this effort is to test a physical activity intervention, for adult clinical care patients at risk of developing cardiovascular disease. The intervention includes 13 weekly and 6 monthly social-cognitive theory-based sessions, remote coaching, a body worn physical activity tracker (PAT), and is delivered online over one year.

A total of n=54 Clinical care patients aged 40-70 years of age with low physical activity (PA) levels (<150 minutes/week) at risk for cardiovascular disease will be recruited. Study outcomes will be measured at baseline, 6 months after intervention start and 12 months after intervention start.

For the primary outcomes, the investigators hypothesize that participants randomized to ActiveGOALSv2 + PAT will have significantly larger (a) increases in step counts/day and % meeting moderate-vigorous physical activity goal of 150 minutes/week (to 12 months) compared to the active PAT control group. Descriptive analyses and graphic displays will be used to identify outliers, missing data, and pattern of attrition. To ensure rigor, the primary analytic strategy will be a linear or generalized mixed-effect models approach in which treatment group, time, and time by group interaction are treated as fixed effects, and subject is treated as a random effect to account for individual subject variability (two sided hypothesis test; .05 level). Mixed models are applicable to longitudinal datasets that contain missing observations, (assuming data is missing at random). Regression modeling will be conducted to adjust for important covariates. The investigators will perform similar analyses to examine changes in secondary outcomes. Descriptive statistics on patient experience, beliefs/attitudes related to maintenance of physical activity changes, and program cost will also be reported.

Power and sample size: For a 2 sided test with alpha level set at .05, and assuming 20% attrition at 12 months, the investigators plan to recruit 54 participants to identify clinically relevant mean difference between randomized groups at 12-months of 2000 steps/day (with a power of .80), and 35% meeting MVPA goal (with a power of .80), given reference mean (sd) values were calculated from baseline waist worn accelerometer data from the current K12 of: 5250 (2200) steps/ day and the investigators assume 5% meeting goal at baseline in the control group.

Descriptive statistics will be used to describe the total eligible population, those referred, and those referred who participated in the study; in order to determine program reach. Exploratory Analysis of Important Pre-Existing Factors: Factor analysis will be used to identify importance of factors related to physical activity levels/ activity goal achievement over the 12 month follow-up (Mplus) from participant EHR data collected prior to intervention start. Factor structures of how individual factors contribute to activity outcomes will be explored at each time point. The best factor structure will be determined with Eigenvalues and fit indices (RMSEA, CFI, and TLI). Factor structures at the 2 time points will be compared at three levels to establish measurement invariance: 1) Configural equivalence, number of factors/ pattern of factor-indicator relationships are identical over time; 2) Metric equivalence, factor loadings are equal over time; and 3) Scalar equivalence, means and values are equivalent over time. Finally, the investigators will use descriptive statistics to report presence/absence of data on physical activity levels, cardiometabolic, and patient-centered outcomes in the EHR. The investigators will apply the same regression approaches utilized in Aim 1a to determine differences between randomized groups for EHR reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-70 years of age
* Low physical activity (PA) levels (<150 minutes/week)
* At least one of the following common cardiometabolic risk factors:

  * high blood pressure:> 129 mm hg SP or >89 mm hg DP or medication
  * high fasting glucose:>100 mg/dl or high HbA1c: ≥42 mmols/mol or medication
  * overweight/ obesity: BMI ≥25 kg/m2).
* Have access to the internet
* Able to read English at a 6th grade level
* Have primary care provider (PCP) permission to increase physical activity without supervision.

Exclusion Criteria:

* Have participated in a physical activity intervention program with behavior tracking and goal setting in the past year.
* Told by a physician that they have diabetes (other than previous gestational diabetes) or have received a diagnosis of cardiovascular disease, regardless of when.
* Pregnant or planning a pregnancy in <12 months
* Non-ambulatory or planning a procedure that will lead to not being ambulatory in <12 months.
* Women who become pregnant during the study will be required to get an updated referral form from their primary care provider (PCP) stating that they are able to increase their physical activity without supervision .

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2022-03-29 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bonny Rockette-Wagner, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled between March 2022 and June 2023.
Pre-assignment Details: Participants were requirement to complete baseline measures for the primary outcome using accelerometer. Participants who withdrew, were found to not be meeting eligibility criteria, or did not completing the measure after consenting were not randomized and were administratively withdrawn.
Period: Overall Study
Arm/Group | PAT (Physical activity monitor) | ActiveGOALSv2
Started | 27 | 27
Completed | 20 | 20
Not Completed | 7 | 7
Not completed — Lost to Follow-up | 6 | 7
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PAT (Physical Activity Monitor) | ActiveGOALSv2 | Total
Number analyzed (Participants) | 27 | 27 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.01 (8.31) | 57.7 (9.26) | 57.36 (8.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 20 | 44
  Male | 3 | 7 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 6 | 12
  White | 19 | 19 | 38
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 27 | 26 | 53
  Unknown or Not Reported | 0 | 0 | 0
Meeting Activity Goal [Count of Participants; unit: Participants] — Based on 150 minutes/week from accelerometer
  Participants | 14 | 17 | 31
Average Moderate-Vigorous Activity [Mean (Standard Deviation); unit: minutes/day] | 29.6 (22.6) | 34.83 (23.48) | 32.3 (23.00)
Average Light Activity [Mean (Standard Deviation); unit: minutes/day] | 338.5 (86.7) | 354.1 (94.1) | 346.5 (90.10)
Average Sedentary [Mean (Standard Deviation); unit: minutes/day] | 455.91 (66.10) | 463.27 (112.57) | 459.65 (91.90)
Average Step Counts [Mean (Standard Deviation); unit: steps/day] | 4564 (2141) | 5023 (2222) | 4797 (2174)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHG] | 122.6 (17.1) | 120.6 (11.9) | 121.6 (14.6)
Body Weight [Mean (Standard Deviation); unit: pounds] | 216.8 (29.9) | 207.4 (33.1) | 212.0 (31.6)
Waist Circumference [Mean (Standard Deviation); unit: centimeters] | 112.8 (16.2) | 108.2 (10.6) | 110.5 (13.7)
Fasting Blood Glucose [Mean (Standard Deviation); unit: mg/dl] | 96.7 (14.5) | 102.6 (16.5) | 99.7 (15.7)
HbA1c [Mean (Standard Deviation); unit: mmol/mol] | 5.42 (0.46) | 5.62 (0.55) | 5.52 (0.52)
LDL Cholesterol [Mean (Standard Deviation); unit: mg/dl] | 116.4 (43.5) | 118.9 (43.4) | 117.6 (43.1)
HDL Cholesterol [Mean (Standard Deviation); unit: mg/dl] | 54.7 (13.0) | 53.0 (15.7) | 53.9 (14.3)
Insulin [Mean (Standard Deviation); unit: mg/dl] | 15.9 (15.1) | 16.0 (10.1) | 16.0 (12.7)
Triglycerides [Mean (Standard Deviation); unit: mg/dl] | 128.9 (54.1) | 162.1 (108.8) | 145.5 (86.7)
Blood Pressure Diastolic [Mean (Standard Deviation); unit: mmHG] | 79 (11) | 79 (9) | 79 (10)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Meeting the Aerobic Activity Goal at 12 Months
Description: Change between 0 and 12 months for y/n meeting the 150 minute/week moderate-vigorous activity goal based on minutes of activity from accelerometer
Time Frame: 12 months versus baseline
Population: Due to participant drop out, incomplete monitor data at 12 months and loss to follow-up there were less people at the 12 month visit with valid monitor data
Measure: Count of Participants; unit: Participants
Arm/Group | PAT (Physical activity monitor) | ActiveGOALSv2
Number analyzed (Participants) | 27 | 27
Participants
  Baseline meeting goal | 11 | 16
  12 months meeting goal: number analyzed (Participants) | 20 | 20
  12 months meeting goal | 11 | 13
Statistical Analysis 1: Comparison: PAT (Physical activity monitor) vs ActiveGOALSv2; Test type: Other; p = 0.63, Mixed Models Analysis — Apriori p-value for significance was <0.05. Models were not adjusted for additional covariates and multiple comparisons adjustment was not performed; Mixed models for binomial outcomes were run to determine if there were significant differences in meeting goal over time

2. Primary Outcome: Change From Baseline in Step Counts at 12 Months
Description: Objectively measured change in step counts between 0 and 12 months using ActiGraph accelerometer
Time Frame: 12 months versus baseline
Population: there were less participants with valid data at the 12 month timepoint due to incomplete monitor data, loss to follow-up, and participant withdraw
Measure: Mean (Standard Error); unit: steps/day
Arm/Group | PAT (Physical activity monitor) | ActiveGOALSv2
Number analyzed (Participants) | 27 | 27
steps/day
  Baseline Adjusted Estimates | 4574.21 (421.86) | 5028.41 (413.78)
  12 month Adjusted Estimates: number analyzed (Participants) | 20 | 20
  12 month Adjusted Estimates | 4533.67 (416.42) | 5680.49 (416.41)
Statistical Analysis 1: Comparison: PAT (Physical activity monitor) vs ActiveGOALSv2; Test type: Other; p = 0.0665, Mixed Models Analysis — Apriori significance level was p<0.05. No adjustment for multiple comparisons was made; Models were not adjusted for additional variables; Mean Difference (Final Values) = -1106.28, Standard Error of Mean 592.76

3. Secondary Outcome: Sedentary Behavior Minutes Over All Timepoints for 12 Months
Description: Objectively measured sedentary behavior over all timepoints for 12 months using ActiGraph accelerometer
Time Frame: 1 week recording; measured at baseline, 6 and 12 months
Reporting Status: Not Posted, anticipated posting 2026-03

4. Secondary Outcome: Moderate-vigorous Activity Minutes Over All Timepoints for 12 Months
Description: Objectively measured moderate-vigorous activity over all timepoints for 12 months using ActiGraph accelerometer
Time Frame: 1 week recording; measured at baseline, 6 and 12 months
Reporting Status: Not Posted, anticipated posting 2026-03

5. Secondary Outcome: Light Activity Minutes Over All Timepoints for 12 Months
Description: Objectively measured Light activity over all timepoints for 12 months using ActiGraph accelerometer
Time Frame: 1 week recording; measured at baseline, 6 and 12 months
Reporting Status: Not Posted, anticipated posting 2026-03

6. Secondary Outcome: Step Counts Over All Timepoints for 12 Months
Description: Objectively measured Step counts over all timepoints for 12 months using ActiGraph accelerometer
Time Frame: 1 week recording; measured at baseline, 6 and 12 months
Reporting Status: Not Posted, anticipated posting 2026-03

7. Secondary Outcome: Patient Experience
Description: patient experience survey designed for this study with the help of patient partners to gather feedback from participants. Feedback will be used in the development of future interventions
Time Frame: measured at 6 and 12 months
Reporting Status: Not Posted, anticipated posting 2026-03

8. Secondary Outcome: Blood Pressure Over All Timepoints for 12 Months
Description: Taken by trained clinic staff using a validated automated blood pressure cuff after participant is seated in an upright position for 5 minutes. Two measure will be taken and the average of the two measures will be used. If the measures are not within 5 mmHG, a third measure will be taken.
Time Frame: measured at baseline, 6 and 12 months
Reporting Status: Not Posted, anticipated posting 2026-03

9. Secondary Outcome: Body Weight Over All Timepoints for 12 Months
Description: will be measured in clinic by trained staff using a validated scale. Participants will be asked to take shoes off and wear light clothes. Average of two measures will be used; if weight is more than .5 pounds different, a third will be taken.
Time Frame: measured at baseline, 6 and 12 months
Reporting Status: Not Posted, anticipated posting 2026-03

10. Secondary Outcome: Waist Circumference Over All Timepoints for 12 Months
Description: will be measured above the iliac crest in clinic by trained staff. Two measures will be taken and averaged; if measures are more than 1 cm different a third measure will be taken.
Time Frame: measured at baseline, 6 and 12 months
Reporting Status: Not Posted, anticipated posting 2026-03

11. Secondary Outcome: Fasting Blood Glucose Over All Timepoints for 12 Months
Description: A fasting blood draw will be taken after 12-16 hours fast.
Time Frame: measured at baseline, 6 and 12 months
Reporting Status: Not Posted, anticipated posting 2026-03

12. Secondary Outcome: HbA1c Over All Timepoints for 12 Months
Description: A fasting blood draw will be taken after 12-16 hours fast.
Time Frame: measured at baseline, 6 and 12 months
Reporting Status: Not Posted, anticipated posting 2026-03

13. Secondary Outcome: LDL Cholesterol Over All Timepoints for 12 Months
Description: A fasting blood draw will be taken after 12-16 hours fast.
Time Frame: measured at baseline, 6 and 12 months
Reporting Status: Not Posted, anticipated posting 2026-03

14. Secondary Outcome: HDL Cholesterol Over All Timepoints for 12 Months
Description: A fasting blood draw will be taken after 12-16 hours fast.
Time Frame: measured at baseline, 6 and 12 months
Reporting Status: Not Posted, anticipated posting 2026-03

15. Secondary Outcome: Perceived Health Score Over All Timepoints for 12 Months
Description: EuroQAL Visual Analogue Scale (EQ-VAS)-Self-reported perception of health on a 0 (lowest possible) to 100 (highest possible) scale.
Time Frame: measured at baseline, 6 and 12 months
Reporting Status: Not Posted, anticipated posting 2026-03

16. Secondary Outcome: Insulin Over All Timepoints for 12 Months
Description: A fasting blood draw will be taken after 12-16 hours fast.
Time Frame: measured at baseline, 6 and 12 months
Reporting Status: Not Posted, anticipated posting 2026-03

17. Secondary Outcome: Triglycerides Over All Timepoints for 12 Months
Description: A fasting blood draw will be taken after 12-16 hours fast.
Time Frame: measured at baseline, 6 and 12 months
Reporting Status: Not Posted, anticipated posting 2026-03

ADVERSE EVENTS:
Time Frame: From enrollment to end of follow-up, 12 months
Arm/Group | PAT (Physical activity monitor) | ActiveGOALSv2
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 0/27 | 0/27

LIMITATIONS AND CAVEATS:
This was a small pilot study that was not powered to assess secondary outcomes. The ability to assess the primary outcome of number of participants meeting goal was affected by several factors including: higher than expected participants meeting goal at baseline (based on accelerometers) and higher than expected non-completion rates for the accelerometers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2025-11-03): https://cdn.clinicaltrials.gov/large-docs/56/NCT04743856/Prot_000.pdf
  • Statistical Analysis Plan (2025-11-03): https://cdn.clinicaltrials.gov/large-docs/56/NCT04743856/SAP_001.pdf
  • Informed Consent Form (2022-02-22): https://cdn.clinicaltrials.gov/large-docs/56/NCT04743856/ICF_002.pdf